CLINICAL TRIAL: NCT07397325
Title: Clinical Study of DA-020 for the Treatment of Chemotherapy Induced Alopecia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Collaborators: Daniel Alain, Inc. (Unknown); Follea International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DA-020-CIA
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chemotherapy Induced Alopecia; Chemotherapy Side Effects
Keywords: Chemotherapy Induced Alopecia; Chemotherapy Alopecia
MeSH Terms: interventions — hyperforin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DA-020 (Active Comparator): Topical DA-020 Solution
  Interventions: Drug: DA-020
- Placebo (Placebo Comparator): Topical Placebo Solution
  Interventions: Drug: Placebo
- DA-020 and Hyperforin (1.5%) (Active Comparator): DA-020 and Hyperforin (1.5%)
  Interventions: Drug: DA-020 and Hyperforin

INTERVENTIONS:
Drug: DA-020 — 7mL application of DA-020 (Topical Oxymetazoline)
  Arms: DA-020
Drug: Placebo — Topical placebo solution
  Arms: Placebo
Drug: DA-020 and Hyperforin — 7mL application of DA-020 (Topical Oxymetazoline) and Hyperforin (1.5%)
  Arms: DA-020 and Hyperforin (1.5%)

SUMMARY:
Clinical Study of DA-020 as a Treatment for Chemotherapy Induced Alopecia

DETAILED DESCRIPTION:
Chemotherapy induced alopecia (CIA) is a common adverse event of oncological treatment. The significant psychological burden of CIA, particularly in women, leads some (~8%) to reject life saving therapeutic regimens. Several studies have demonstrated the effectiveness of scalp vasoconstriction as a prophylactic treatment for CIA. Recently, US Food and Drug Administration (FDA) approved a scalp-cooling device as a prophylactic treatment for CIA. Scalp cooling results in reduced local blood perfusion and consequently reduced chemotherapeutic agents reaching the hair follicle niche; however, scalp cooling requires prolongation of the time required to attend the chemotherapy unit (>2 hrs) as well as common adverse events including intolerance to cold. A previous study demonstrated that the α1 agonist, phenylephrine hydrochloride, applied topically can penetrate the scalp and bind α1 receptors. As such, a topically applied α1 agonist would reduce scalp blood perfusion. A novel formula (DA-020), containing an α1 agonist, that can also penetrate the scalp and bind α1 receptors. The aim of the study is to test the hypothesis that DA-020 can reduce scalp blood perfusion and thus reduce hair loss due to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage I or stage II breast cancer
* Scheduled but not begun, at least 4 cycles of taxane and/or anthracycline-based chemotherapy.
* Ages 18-65
* Able to give informed consent

Exclusion Criteria:

* Resting blood pressure outside the range of 105-140/ 55-99
* Uncontrolled or severe hypertension
* Female pattern hair loss or hair loss disorder
* Folliculitis
* Scalp psoriasis
* Seborrheic dermatitis
* Inflammatory scalp conditions such as lichen planopillaris
* Subjects wearing wigs prior to chemotherapy
* Use of MAO inhibitors
* Unable to provide consent or make allotted clinical visits

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2026-03-16 (Estimated); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
Prevention of Hair Loss (Common Terminology Criteria for Adverse Events V5.0) | Week [0,12]
  Amount of hair loss during chemotherapy treatment measured by the Common Terminology Criteria for Adverse Events (CTCAE) V5.0. The Common Terminology Criteria for Adverse Events is a common terminology developed by the National Cancer Institute to describe and grade adverse events related to cancer therapy.

SECONDARY OUTCOMES:
Hair Re-Growth Post Treatment (Common Terminology Criteria for Adverse Events V5.0) | Week [12, 24]
  Amount of hair re-growth post chemotherapy treatment measured by the Common Terminology Criteria for Adverse Events (CTCAE) V5.0. The Common Terminology Criteria for Adverse Events is a common terminology developed by the National Cancer Institute to describe and grade adverse events related to cancer therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Goren, MD, Study Director — University of Rome G. Marconi
Locations (1):
- University of Rome ("G. Marconi"), Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fahl WE. Complete prevention of radiation-induced dermatitis using topical adrenergic vasoconstrictors. Arch Dermatol Res. 2016 Dec;308(10):751-757. doi: 10.1007/s00403-016-1691-2. Epub 2016 Oct 4. PMID 27704205
- [Background] Soref CM, Fahl WE. A new strategy to prevent chemotherapy and radiotherapy-induced alopecia using topically applied vasoconstrictor. Int J Cancer. 2015 Jan 1;136(1):195-203. doi: 10.1002/ijc.28961. Epub 2014 May 16. PMID 24811525